CLINICAL TRIAL: NCT04470986
Title: International Registry on the Diagnosis and Treatment of Inferior Vena Cava Thrombosis
Brief Title: Study on Inferior Vena Cava Thrombosis
Acronym: SIVECT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: International Society on Thrombosis and Haemostasis (Unknown)
Responsible Party: Principal Investigator, Dr. Omri Cohen, Unusual site thrombosis service, Sheba Medical Center
Other Study IDs: SHEBA-20-7345-OC-CTIL
Record Dates: First submitted 2020-07-08; First posted 2020-07-14 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Inferior Vena Cava Thrombosis
Keywords: Inferior vena cava (IVC); Thrombosis; Anticoagulation; Deep vein thrombosis (DVT)
MeSH Terms: conditions — Thrombosis; Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will focus on patients having inferior vena cava (IVC) thrombosis, either with or without thrombosis in other veins.

The purpose of this study is to assess risk factors, safety and effectiveness of treatment options, and outcomes of patients with IVC thrombosis.

DETAILED DESCRIPTION:
Thrombosis of the inferior vena cava (IVC) is a rare form of deep venous thrombosis (DVT). Optimal treatment strategies and clinical outcomes are not well established.

This multicenter, international, observational study will assess the effectiveness and safety of current treatment options in patients with IVC thrombosis, and describe the long-term outcomes of patients with IVC thrombosis.

Patients with an objective diagnosis of IVC thrombosis, either with or without proximal lower extremity DVT will be included. Information will be collected on baseline characteristics, risk factors for thrombosis, symptoms, mode of diagnosis, presence of concomitant lower limb DVT, PE, IVC filter or unusual site thrombosis (splanchnic, gonadal and renal veins), treatment modalities (anticoagulation and/or thrombolysis), choice of anticoagulant, dose and duration of treatment, recanalization assessment (if available), recurrence of VTE during follow up, bleeding according to International Society on Thrombosis and Haemostasis criteria, development post-thrombotic syndrome (PTS) according to Villalta score and mortality during follow up. Patients should be followed up for 24 months from diagnosis. The number of visits is left to the discretion of the treating physician, but information on clinical outcomes at two intermediate time points is requested.

ELIGIBILITY:
Inclusion criteria:

1. Consecutive adult patients (> 18 years) with an objective diagnosis of IVC thrombosis, either with or without proximal lower extremity DVT (involving the femoral, common femoral, or iliac veins) will be eligible for the study.
2. Diagnosis should be obtained by either doppler ultrasonography, CT angiography or MRI angiography.
3. Patients who had objective diagnosis of IVC thrombosis within 6 months prior to the starting of the registry will also be eligible, providing they are prospectively followed up by the participating centers and all requested information is available.

Exclusion criteria:

Patients enrolled in interventional studies.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with an objective diagnosis of IVC thrombosis, either with or without proximal lower extremity DVT
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Rates of venous thromboembolism (VTE) recurrence | 2 Years
  Recurrence of any venous thrombosis (not previously diagnosed)
Rate of all cause mortality | 2 Years
  Mortality (patient's death) from any cause
Rates of major bleeding | 2 Years
  Major bleeding per International Society on Thrombosis and Haemostasis criteria Schulman S, Kearon C, Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of major bleeding in clinical investigations of antihemostatic medicinal products in non-surgical patients. J Thromb Haemost 2005; 3: 692- 4.

SECONDARY OUTCOMES:
Rates of thrombosis recanalization | 2 Years
  Evidence of thrombosis resolution by imaging (none/partial/complete, with regard to the latest imaging study), with time from initiation of therapy to thrombus resolution being calculated accordingly.
Rates of post-thrombotic syndrome (PTS) | 2 Years
  According to:
  Goldenberg NA, Brandão L, Journeycake J, Kahn S, Monagle P et al. Definition of post-thrombotic syndrome following lower extremity deep venous thrombosis and standardization of outcome measurement in pediatric clinical investigations. J Thromb Haemost. 2012 Mar;10(3):477-80.
Rates of clinically relevant non-major bleeding | 2 Years
  Clinically relevant non-major bleeding per International Society on Thrombosis and Haemostasis criteria Kaatz S, Ahmad D, Spyropoulos AC, Schulman S, Subcommittee on Control of Anticoagulation of the Scientific and Standardization Committee of the International Society on Thrombosis and Haemostasis. Definition of clinically relevant non-major bleeding in studies of anticoagulants in atrial fibrillation and venous thromboembolic disease in non-surgical patients: communication from the SSC of the ISTH. J Thromb Haemost. 2015 Nov;13(11):2119-26.

IPD SHARING:
Plan to Share IPD: Undecided